CLINICAL TRIAL: NCT05622474
Title: A Multicenter Randomized Controlled Clinical Study on the Treatment of T3N1M0 High Risk Nasopharyngeal Carcinoma With or Without Induction Chemotherapy Before Concurrent Radiotherapy and Chemotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2022-589
Record Dates: First submitted 2022-11-13; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; T3N1M0; Induction Chemotherapy; Concurrent Chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Induction Chemotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IC plus CC plus IMRT (Experimental): Induction chemotherapy followed by Intensity-modulated radiotherapy plus concurrent chemotherapy
  Interventions: Drug: Induction chemotherapy plus Concurrent chemotherapy; Radiation: IMRT
- CC plus IMRT (Active Comparator): Intensity-modulated radiotherapy plus concurrent chemotherapy alone
  Interventions: Drug: Concurrent chemotherapy; Radiation: IMRT

INTERVENTIONS:
Drug: Induction chemotherapy plus Concurrent chemotherapy — Induction chemotherapy: TP( Docetaxel 75mg/m2, D1 and cisplatin 25 mg/m2, D1-3 every 3 weeks for 3 cycles) OR GP (Gemcitabine 1000mg/m2，D1,D8 and cisplatin 25 mg/m2, D1-3 every 3 weeks for 3 cycles）
  Concurrent chemotherapy: DDP -- Cisplatin 25 mg/m2, D1-3 , every 3 weeks for 2 cycles during radiation.
  Arms: IC plus CC plus IMRT
Drug: Concurrent chemotherapy — Concurrent chemotherapy: DDP -- Cisplatin 25 mg/m2, D1-3 , every 3 weeks for 2 cycles during radiation.
  Arms: CC plus IMRT
Radiation: IMRT — Radical radiation: Intensity-modulated radiotherapy

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of curative radiotherapy with or without induction chemotherapy in patients with T3N1M0 nasopharyngeal carcinoma. The main question[s] it aims to answer are:

* Whether induction chemotherapy confers a survival benefit in patients with T3N1M0 nasopharyngeal carcinoma with high risks factors.
* Whether induction chemotherapy worsens adverse effects in patients with T3N1M0 nasopharyngeal carcinoma.

Participants in experimental group will receive 3 cycles induction chemotherapy (GP or TPF) followed by concurrent chemoradiotherapy.Participants in control group will receive concurrent chemoradiotherapy only.

Researchers will compare FFS, OS and AE or SAE to see if patients can benefit from induction chemotherapy or screen out high-risk factors associated with survival benefits.

DETAILED DESCRIPTION:
In this study, 236 patients with pathologically diagnosed nasopharyngeal carcinoma and clinical stage of T3N1M0 will be randomly divided into two groups, 118 in the experimental group (induction chemotherapy + concurrent chemoradiotherapy) and 118 in the control group (concurrent chemoradiotherapy). The experimental group received 3 courses of induction chemotherapy followed by radical radiotherapy for the nasopharynx and neck, and 2-3 courses of cisplatin (100mg/m2, Q3W) treatment during radiotherapy. The control group received radical radiotherapy for the nasopharynx and neck, and 2-3 courses of cisplatin (100mg/m2, Q3W) during radiotherapy. Since there have been clinical trials to prove that GP or TPF induction chemotherapy is effective in locally advanced nasopharyngeal carcinoma, the induction chemotherapy regimen in this study can be selected by the investigator with GP or TPF. During treatment and within 3 years after treatment, the efficacy and safety of patients in both groups were followed up and evaluated.

ELIGIBILITY:
Inclusion Criteria:

1.Pathologically diagnosed with stage T3N1M0 nasopharyngeal cancer according to 2017 AJCC Cancer Staging Manual-8th Edition; not received anticancer treatment.

2.18-70 years old. 3. One or more of the following prognostic factors exist:

1. MRI showed extravasation of lymph node capsule,
2. MRI showed lymph node necrosis,
3. The maximum diameter of positive lymph nodes in the three-dimensional direction on MRI is ≥ 3cm,
4. 2 or more positive lymph nodes,
5. Peripheral blood EBV-DNA ≥ 4000 copies/ml,
6. The maximum SUV value of lymph nodes on PET/CT ≥ 9.3. 4.ECOG Score (PS score) 0 or 1. 5.Neutrophil count > 1.5*10^9/L, hemoglobin > 90g/L, and platelet count > 100*10^9/L.

6.ALT or AST level < 2.5 times upper normal limit (upper limit of normal, ULN), bilirubin level < 1.5 times ULN.

7.Creatinine clearance level > 60 ml/min. (Calculated according to Cockcroft Gault formula).

8.Patients must sign an informed consent and must be willing and able to comply with the visit, treatment protocol, laboratory tests and other requirements specified in the study protocol.

Exclusion Criteria:

1. Patients who have other malignant tumors within 5 years, excluding carcinoma in situ, well treated non melanoma skin cancer and papillary thyroid cancer.
2. Other conditions that may affect the safety or test compliance of the subject as judged by the investigator, including symptomatic heart failure, unstable angina, myocardial infarction, active infection requiring systemic treatment, mental illness or family and social factors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Failure Free Survival | Two years
  The absence of relapse, non-relapse mortality or addition of another systemic therapythe last follow-up if there is no disease progression.

SECONDARY OUTCOMES:
Overall survial | Two years
  The time from randomization until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Fang-Yun Xie, M.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No